CLINICAL TRIAL: NCT00355992
Title: The Ischemia Modified Albumin In Diagnosing Ischemic New Events (IMAGINE Study).
Brief Title: The Ischemia Modified Albumin In Diagnosing Ischemic New Events
Acronym: IMAgine
Status: Terminated | Type: Observational
Sponsor: Inverness Medical Innovations (Industry)
Responsible Party: Bob Parson, Inverness Medical Innovations
Other Study IDs: IMA-0106-001.04
Record Dates: First submitted 2006-06-27; First posted 2006-07-25 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-05

CONDITIONS: Heart Disease, Ischemic; Ischemia, Myocardial; Ischemic Heart Disease; Unstable Angina
Keywords: Myocardial Ischemia; Chest pain; Ischemia Modified Albumin; Acute Coronary Syndrome
MeSH Terms: conditions — Myocardial Ischemia; Angina, Unstable; Chest Pain; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of the study is to evaluate the utility of Ischemia Modified Albumin (IMA) for risk stratification in patients presenting with chest discomfort and possible ischemic heart disease, and to evaluate the diagnostic and prognostic implication for IMA for major adverse cardiac events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary complaints of chest discomfort or patients with symptoms indicative of a moderate to high probability for unstable angina clinically indicated reason for evaluation for ACS in the Emergency Department meeting tyhe following inclusion criteria will be enrolled:
* Age >=21 years
* Presentation within two hours of relief of most recent episode of chest pain or presence of on-going symptoms suggestive of coronary ischemia, which should be at least 10 minutes in duration.
* Patients being evaluated for suspected ischemic signs and or symptoms (chest pain) at the time of presentation according to routine standard of care institutional chest pain protocol/pathway.

Exclusion Criteria:

* Administration of thrombolytic medication prior to first (presentation) blood draw
* Acute coronary syndrome (ACS) secondary to supply/demand inequity (i.e. known anemia, tachycardia, - defined as HR greater than 150 bpm, known sepsis, hypotension, defined as blood pressure < 90 mmHg).
* Established diagnosis of liver cirrhosis
* Other acute ischemic sources (ongoing severe claudication, mesenteric ischemia, acute TIA/CVA)
* Renal failure requiring dialysis
* Greater than 2 hours from relief of the most recent episode of chest pain or signs and symptoms suggestive of coronary ischemia.
* Chest pain following traumatic injury to the chest
* Evidence for sever systemic infection, manifesting as fever (temperature >100 degrees) and systolic blood pressure <100 mmHg
* Patients unwilling or unable to provide written consent, without available next of kin
* Cocaine-related chest pain
* Pregnancy
* Known diagnosis of active malignancy
* Acute Bowel Ischemia
* Severe peripheral vascular disease
* Acute brain ischemia

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present in the emergency department at the listed institutions with suspected ischemic signs and or symptoms (chest pain) will be eligible for participation in the study as long as they meet inclusion and exclusion criteria and sign an informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2006-09; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: James L Januzzi, M.D., Study Director — Massachusetts General Hospital
Locations (5):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dartmouth Medical Center, Lebanon, New Hampshire
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University, Nashville, Tennessee
- Hamilton General Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Bhardwaj A, Truong QA, Peacock WF, Yeo KT, Storrow A, Thomas S, Curtis KM, Foote RS, Lee HK, Miller KF, Januzzi JL Jr. A multicenter comparison of established and emerging cardiac biomarkers for the diagnostic evaluation of chest pain in the emergency department. Am Heart J. 2011 Aug;162(2):276-282.e1. doi: 10.1016/j.ahj.2011.05.022. PMID 21835288